CLINICAL TRIAL: NCT06416345
Title: Cue2Walk, Cost-effectiveness of Automated Freezing Detection and Provision of External Cues in Comparison to Usual Care in People With Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Erwin E. H. van Wegen, Principal Investigator, Associate Professor Neurorehabilitation, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL86310.018.24
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Freezing of Gait; (Smart) Cueing; Costeffectiveness
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): At-home use of the Cue2Walk
  Interventions: Device: Cue2Walk
- Control Group (Other): Usual Care (+ Waiting List)
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Cue2Walk — 24 weeks of using of the Cue2Walk device in the own living environment + 8 weeks of naturalistic follow-up
  Arms: Intervention Group
Other: Usual Care — 24 weeks of receiving usual care + 8 weeks of using of the Cue2Walk device in the own living environment
  Arms: Control Group

SUMMARY:
The majority of people with Parkinson's disease incur Freezing of Gait (FoG), which is not addressed adequately by medication. Cueing is a proven strategy to overcome FoG. The Cue2Walk is a device with automated detection of FoG and provision of rhythmic cues. In this study, the (cost-)effectiveness of the Cue2Walk device as compared to usual care is investigated.

DETAILED DESCRIPTION:
Freezing of gait (FoG) is one of the most common and disabling motor symptoms of Parkinson's disease and is associated with poorer quality of life. However, current pharmacological or even surgical treatments do not address FoG adequately and innovative rehabilitation strategies are needed. Cueing is a proven strategy to overcome FoG episodes and an essential part in the management of FoG. The Cue2Walk, a Medical Device Class I CE-certified leg-worn device, addresses the debilitating effects of FoG episodes at home with 'smart cueing' by combining automatic detection of a freezing episode with manual or automatic rhythmic cues (auditory or vibro-tactile). This study aims to investigate the (cost-)effectiveness of the Cue2Walk device as compared to usual care. This study is a multicenter randomized clinical trial with 2 parallel groups (24-week intervention group and 24-week 'waiting list' group). After 24 weeks, an 8-week naturalistic follow-up will be implemented for the intervention group, while participants in the waiting list group will also receive the intervention, but for 8 weeks. Frequently repeated assessment of outcomes measures will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease according to UK Brain bank criteria
* Daily Freezing of Gait
* Hoehn-Yahr stage 2-4
* Stable medication regime and/or DBS settings as determined by the treating neurologist
* Ability to walk 5 minutes while unassisted by another person

Exclusion Criteria:

* Participation in another clinical study
* Use of a personal cueing device at home
* Previous use of the Cue2Walk medical device
* Presence of co-morbidities that would hamper participation
* Cognitive impairment preventing understanding of therapeutic instructions (Montreal Cognitive Assessment (MoCA) Score <16)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported quality of life | Baseline (week 0), week 8, week 16, Post-intervention (week 24), week 32
  Self-reported quality of life will be determined using the Parkinson's Disease Questionnaire (PDQ-39)
General health-related quality of life | Baseline (week 0), week 8, week 16, Post-intervention (week 24), week 32
  General health-related quality of life will be determined using the EuroQol 5 Dimensions 5 Level Survey (EQ-5D-5L)
Time in Freezing of Gait | Continuously from baseline (week 0) up to week 32
  Time in Freezing of Gait (i.e. frequency and duration of FoG) will be determined by the Cue2Walk medical device

SECONDARY OUTCOMES:
Falls Efficacy | Baseline (week 0), week 8, week 16, Post-intervention (week 24), week 32
  The level of concern about falling during various activities will be determined by the Falls Efficacy Scale International (FES-I)
Numbers of falls | Weekly from baseline (week 0) up to week 32
  The number of falls and near-falls will be determined with a weekly diary
Freezing of Gait severity | Baseline (week 0), week 8, week 16, Post-intervention (week 24), week 32
  Freezing of Gait severity will be determined by the New Freezing of Gait Questionnaire (NFOG-Q)
Freezing of Gait severity | Baseline (week 0), week 8, week 16, Post-intervention (week 24), week 32
  Freezing of Gait severity will be determined by the Patient Reported Outcomes for Freezing of Gait (PRO-FOG)
Independence in Activities of Daily Living | Baseline (week 0), week 8, week 16, Post-intervention (week 24), week 32
  Independence in Activities of Daily Living will be determined by the Nottingham Extended Activities of Daily Living Index (NEADL)
Motor Aspects of Experiences of Daily Living | Baseline (week 0), week 8, week 16, Post-intervention (week 24), week 32
  Motor Aspects of Experiences of Daily Living will be determined by MDS-UPDRS part II
Daily mobility | Continuously from baseline (week 0) up to week 32
  Daily mobility will be determined by the Cue2Walk step count
Mood | Baseline (week 0), week 8, week 16, Post-intervention (week 24), week 32
  Mood will be determined by Hospital Anxiety and Depression Scale (HADS)
Gait-Specific Attentional Profile | Baseline (week 0), week 8, week 16, Post-intervention (week 24), week 32
  Gait-Specific Attentional Profile will be determined by the Gait-Specific Attentional Profile questionnaire (G-SAP)
Acceptance of Illness | Baseline (week 0), week 8, week 16, Post-intervention (week 24), week 32
  Acceptance of illness will be determined by the Chronic Illness Acceptance Questionnaire (CIAQ)
Caregiver burden | Baseline (week 0), week 8, week 16, Post-intervention (week 24), week 32
  Caregiver burden will be determined by Zarit's Burden Interview Short Form (ZBI-12)
Patient experiences | Baseline (week 0), week 8, week 16, Post-intervention (week 24), week 32
  We will use patient reported experience measures (PREMS) to quantify patient experiences regarding the care they receive during the intervention phase and we will record user experiences

OTHER OUTCOMES:
Resource Utilization | Baseline (week 0), week 8, week 16, Post-intervention (week 24)
  For the economic evaluation, resource utilization will be determined by a cost questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Erwin EH van Wegen, Dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands